CLINICAL TRIAL: NCT00720473
Title: Lamotrigine Therapy in the Treatment of Geriatric Bipolar Depression: An Evaluation of Markers of Cerebral Energy Metabolism
Brief Title: Lamotrigine Therapy in Geriatric Bipolar Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mclean Hospital (Other)
Responsible Party: Principal Investigator, Brent Forester, Director, Mood Disorders Division, Geriatric Psychiatry Research Program, Mclean Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2005-P-002493
Record Dates: First submitted 2008-07-18; First posted 2008-07-22 (Estimated); Results first posted 2016-07-21 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Bipolar Depression
Keywords: Bipolar depression; Elderly; Lamotrigine; Brain energy metabolism
MeSH Terms: conditions — Bipolar Disorder | interventions — Lamotrigine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A: Other (Other): Open Label Study
  Interventions: Drug: Lamotrigine
- B: Healthy Controls (No Intervention)

INTERVENTIONS:
Drug: Lamotrigine — Lamotrigine with dosage range from 25 mg to 200 mg per day.
  Other Names: Lamictal
  Arms: A: Other

SUMMARY:
We propose to study the efficacy and tolerability of lamotrigine in the treatment of older adults with bipolar depression and to compare measures of brain energy metabolism between older subjects with bipolar depression and healthy age-matched controls in order to better understand treatment response in geriatric bipolar depression.

DETAILED DESCRIPTION:
We will use MRI techniques and neuropsychological testing to investigate potential markers of treatment response in elderly bipolar depressed patients receiving lamotrigine and age-matched, non-depressed controls.

We intend to test these hypotheses:

1. At least 50% of older subjects with bipolar depression will respond treatment with lamotrigine as evidenced by a 50% reduction on the Montgomery Asberg Rating Scale (MADRS). In addition, treatment with lamotrigine will be safe and well tolerated as evidenced by a drop-out rate of less than 10% due to adverse effects.
2. Compared with healthy age-matched, non-demented, non-depressed controls, subjects with geriatric bipolar depression will demonstrate abnormalities in cerebral energy metabolism as assessed by elevated levels of glutamate and lactate, and decreased levels of NAA, using 1H MRS at 4T.
3. Successful treatment with lamotrigine in geriatric bipolar depression will result in decreases in lactate and glutamate, and elevations in NAA.
4. Baseline measures of executive functioning and information processing speed (measured by performance on the Wisconsin Card Sorting Test (WCST), Trails A and B and Stroop tests) will be impaired in subjects with geriatric bipolar depression compared with healthy controls. These measures will improve with successful treatment with lamotrigine and correlate with improvements in markers of cerebral energy metabolism (lactate, glutamate, NAA).

ELIGIBILITY:
Inclusion Criteria (for Bipolar Subjects):

* 60 years or older
* Meet DSM-IV diagnostic criteria for Bipolar Disorder, Current Episode Depressed
* First episode of mania before the age of 50 (early-onset bipolar disorder)
* Montgomery-Asberg Depression Rating Scale (MADRS) Score of greater or equal to 20.
* Young Mania Rating Scale (YMRS) of less than or equal to 6.
* Able to provide informed consent
* Must speak English
* Must be able to visit McLean Hospital for the screening visit and six study visits during the 8-week duration of the study.
* Subjects may be taking other medications for bipolar depression including antidepressants, mood stabilizers and antipsychotic mediations prior to lamotrigine therapy, but may not have any dosage adjustments of these medications in the week before lamotrigine is added.

Exclusion Criteria (for Bipolar Subjects):

* Serious or unstable medical illness, including cardiovascular, hepatic, renal, respiratory, endocrine, neurologic or hematologic disease.
* History of seizure disorder
* History or current diagnosis of the following psychiatric illnesses: any organic mental disorder (including dementia), schizophrenia, schizoaffective disorder, delusional disorder, psychotic disorder not otherwise specified, unipolar major depressive disorder, patients with substance dependence disorders, including alcohol, active within the last 12 months.
* First episode of mania after the age of 50 (to exclude late-onset bipolar disorder)
* History of multiple adverse drug reactions or allergy to the study drugs.
* Use of medications that are excluded in this study (benzodiazepines, barbiturates; however, the use of non-benzodiazepine sedative hypnotics (such as zolpidem (Ambien)) may be used as needed except within 48 hours of the MRI scan)
* Any of the exclusion criteria mentioned in the MRI risks section below

Inclusion Criteria (for Controls):

* 60 years or older
* Able to provide informed consent
* Must speak English
* Women entering this study must be post-menopausal

Exclusion Criteria (for Controls):

- Same criteria for the Bipolar Depressed group with the exception of the "first episode of mania" which is not applicable.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2006-04; Primary Completion 2011-07 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brent P Forester, MD, Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- A: BPD Subjects: Open Label Study
  Lamotrigine : Lamotrigine with dosage range from 25 mg to 200 mg per day.
- B: Healthy Control: No Intervention
Period: Overall Study
Arm/Group | A: BPD Subjects | B: Healthy Control
Started | 45 | 24
Completed | 15 | 16
Not Completed | 30 | 8

BASELINE CHARACTERISTICS:
Population: Baseline scans were available for 37 participants, 23 BPD subjects and 14 for healthy controls. One participant had missing scan data, and twenty one participants with a BPD diagnosis had baseline MADRS scores available.
Groups:
- BPD Subjects: Open Label Study
  Lamotrigine : Lamotrigine with dosage range from 25 mg to 200 mg per day.
- Control Subjects: Age matched controls without BPD
- Total: Total of all reporting groups
Arm/Group | BPD Subjects | Control Subjects | Total
Number analyzed (Participants) | 23 | 14 | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 7 | 24
  >=65 years | 6 | 7 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.0 (5.9) | 67.5 (8.8) | 64.6 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 16
  Male | 14 | 7 | 21
Region of Enrollment [Number; unit: participants]
  United States | 23 | 14 | 37

OUTCOME MEASURES:

1. Primary Outcome: Mean Glutamine to Creatine Ratio by Diagnosis at Baseline
Time Frame: Baseline
Population: Baseline scans were available for 37 participants. One participant was missing scan data.
Measure: Mean (Standard Deviation); unit: mean serum Glutamine to Creatine ratio
Arm/Group | BPD Subjects | Control Subjects
Number analyzed (Participants) | 22 | 14
mean serum Glutamine to Creatine ratio | .34 (.12) | .36 (.18)

2. Primary Outcome: Mean Glutamate to Creatine Ratio by Diagnosis at Baseline
Time Frame: Baseline
Population: Baseline scans were available for 37 participants. One participant was missing scan data.
Measure: Mean (Standard Deviation); unit: mean serum Glutamate to Creatine ratio
Arm/Group | BPD Subjects | Control Subjects
Number analyzed (Participants) | 22 | 14
mean serum Glutamate to Creatine ratio | .96 (.29) | .85 (.25)

3. Primary Outcome: Mean N-Acetyl Aspartate (NAA) to Creatine Ratio by Diagnosis at Baseline
Time Frame: Baseline
Population: Baseline scans were available for 37 participants. One participant was missing scan data.
Measure: Mean (Standard Deviation); unit: Mean NAA to creatine ratio
Arm/Group | BPD Subjects | Control Subjects
Number analyzed (Participants) | 22 | 14
Mean NAA to creatine ratio | 0.97 (0.14) | 0.84 (0.22)

4. Primary Outcome: Associations Between Depression Symptom Severity and Glutamate to Creatine Ratio at Baseline
Description: Estimated changes in least squares mean in the metabolite ratio per 10-point increase in MADRS score. The minimum MADRS score is 0 and the maximum is 60, with 60 being the most depressed. Estimate was from linear regression models controlling for age and sex. The change is across regions, parieto-occipital and anterior cingulate cortex.
Time Frame: Baseline
Population: Association between depression symptom severity and metabolite ratios were only conducted in the depressed group, because there should be no change in MADRS score for non-depressed control subjects who received no treatment.
Measure: Least Squares Mean (95% Confidence Interval); unit: Glu:Cr/+10 MADRS
Groups:
- A: Other: Open Label Study
  Lamotrigine : Lamotrigine with dosage range from 25 mg to 200 mg per day.
Arm/Group | A: Other
Number analyzed (Participants) | 21
Glu:Cr/+10 MADRS | 0.18 [-0.02 to 0.38]

5. Primary Outcome: Estimated Change in Least Squares Mean in Glutamate to Creatine Ratio Between Baseline and Follow-up
Description: Follow-up Least Squares Mean - Baseline Least Squares Mean
Time Frame: 8 Weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: serum Glutamate to Creatine ratio
Arm/Group | BPD Subjects | Control Subjects
Number analyzed (Participants) | 13 | 11
serum Glutamate to Creatine ratio | 0.00 [-0.17 to 0.16] | -0.12 [-0.30 to 0.07]

6. Primary Outcome: Estimated Change in Least Squares Mean in the Glutamine to Creatine Ratio Between Baseline and Follow-up
Description: Follow-up Least Squares Mean - Baseline Least Squares Mean
Time Frame: 8 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: serum Glutamine to Creatine ratio
Arm/Group | BPD Subjects | Control Subjects
Number analyzed (Participants) | 13 | 11
serum Glutamine to Creatine ratio | 0.02 [-0.09 to 0.14] | 0.08 [-0.05 to 0.21]

7. Primary Outcome: Estimated Change in Least Squares Mean in the NAA to Creatine Ratio Between Baseline and Follow-up
Description: Follow-up Least Squares Mean - Baseline Least Squares Mean
Time Frame: 8 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: NAA to creatine ratio
Arm/Group | BPD Subjects | Control Subjects
Number analyzed (Participants) | 13 | 11
NAA to creatine ratio | 0.06 [-0.06 to 0.19] | -0.03 [-0.16 to 0.10]

8. Primary Outcome: Association of MADRS Changes With Glutamate to Creatine Ratio Changes From Baseline to Follow-up
Description: Estimated least squares mean metabolite ratio changes with a 10-point decrease in MADRS score. The MADRS minimum score is 0 and maximum is 60, with 60 being the most depressed score. Estimate was from linear regression models controlling for age and sex. The change is across regions, parieto-occipital and anterior cingulate cortex.
Time Frame: 8 Weeks
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: Glu:Cr/-10 MADRS
Arm/Group | BPD Subjects
Number analyzed (Participants) | 11
Glu:Cr/-10 MADRS | -.007 [-0.24 to 0.23]

9. Primary Outcome: Associations of MADRS Changes With Glutamine to Creatine Ratio Changes From Baseline to Follow-up
Description: Estimated least squares mean metabolite ratio changes with a 10-point decrease in MADRS score. MADRS minimum score is 0 and maximum is 60, with 60 being most depressed. Estimate was from linear regression models controlling for age and sex. The change is across regions, parieto-occipital and anterior cingulate cortex.
Time Frame: 8 weeks
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: Gln:Cr/-10 MADRS Score
Arm/Group | BPD Subjects
Number analyzed (Participants) | 11
Gln:Cr/-10 MADRS Score | 0.04 [-0.07 to 0.14]

10. Primary Outcome: Associations of MADRS Changes With NAA to Creatine Ratio Changes From Baseline to Follow-up
Description: as for outcome 9
Time Frame: 8 weeks
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: NAA:Cr/-10 MADRS
Arm/Group | BPD Subjects
Number analyzed (Participants) | 11
NAA:Cr/-10 MADRS | 0.05 [-0.04 to 0.15]

11. Primary Outcome: Mean Montgomery Asberg Depression Rating Scale (MADRS) Score at Baseline
Description: The minimum MADRS score is 0 and the maximum is 60, with 60 being the most depressed.
Time Frame: Baseline
Population: MADRS scores were available for 27 eligible bipolar subjects and 14 eligible controls.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BPD Subjects | Control Subjects
Number analyzed (Participants) | 27 | 14
units on a scale | 24.78 (6.65) | 1.03 (1.55)

12. Primary Outcome: Means of MADRS Scores at 8 Weeks
Description: The minimum MADRS score is 0 and the maximum is 60, with 60 being the most depressed.
Time Frame: 8 Weeks
Population: MADRS scores were available for 16 bipolar subjects who completed the protocol and 8 healthy controls.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BPD Subjects | Control Subjects
Number analyzed (Participants) | 16 | 8
units on a scale | 18.31 (9.41) | 1.38 (1.51)

ADVERSE EVENTS:
Arm/Group | Control Subjects | BPD Subjects
Serious Adverse Events (participants affected / at risk) | 0/24 | 2/45
Other Adverse Events (participants affected / at risk) | 0/24 | 14/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Subjects (N=24) | BPD Subjects (N=45)
Loss of consciousness (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Subject fell off bicycle and lost consciousness.
Mania (Psychiatric disorders) | 0 (0) | 1 (1) — Subject was hospitalized due to mania
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Subjects (N=24) | BPD Subjects (N=45)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Subject developed a rash, which was found to be unrelated by the subject's dermatologist.
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Subject developed a rash after taking second dose.
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Subject reported developing a blister on the hand.
mania (Psychiatric disorders) | 0 (0) | 1 (1) — Subject entered a manic state, with decreased sleep, pressured speech, and delusions.
Blurry Vision (Eye disorders) | 0 (0) | 1 (1) — Subject reported blurry vision
Insomnia (Psychiatric disorders) | 0 (0) | 4 (4) — Four subjects reported sleep disturbances.
Decreased balance (General disorders) | 0 (0) | 3 (3) — Three subjects reported feeling unbalanced or dizzy.
Stomach upset (Gastrointestinal disorders) | 0 (0) | 2 (2) — Two subject reported gastrointestinal problems including upset stomach and indigestion.
Irritability (Psychiatric disorders) | 0 (0) | 1 (1) — One subject experienced increased irritability
Headache (General disorders) | 0 (0) | 2 (2) — Two subjects reported mild headaches.
Runny Nose (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — One subject reported a mild runny nose.
Weight gain (Metabolism and nutrition disorders) | 0 (0) | 1 (1) — A subject reported gaining one pound.

LIMITATIONS AND CAVEATS:
Limited data was available for associating changes in MADRS scores with metabolite changes (22 regions from 11 participants with BPD).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No